CLINICAL TRIAL: NCT06176963
Title: An Open-label, Single Group, Single-dose Clinical Study to Evaluate the Usability of the Pre-filled Syringe of SB11 in Subjects With Neovascular Age-Related Macular Degeneration or Macular Oedema Secondary to Retinal Vein Occlusion
Brief Title: A Study to Evaluate the Usability of the SB11 PFS in Subjects With Wet AMD or Macular Oedema Secondary to RVO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Bioepis Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SB11-2001
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Results first posted 2024-12-30 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Neovascular Age-related Macular Degeneration; Macular Edema; Retinal Vein Occlusion
MeSH Terms: conditions — Macular Edema; Retinal Vein Occlusion | interventions — Ranibizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- SB11 PFS (Experimental): Subjects received a single dose of SB11 PFS containing 0.5 mg ranibizumab in 0.05 mL solution.
  Interventions: Combination Product: SB11 PFS

INTERVENTIONS:
Combination Product: SB11 PFS — SB11 provided in a pre-filled syringe (PFS) containing 0.5 mg ranibizumab in 0.05 mL for ITV injection
  Other Names: Ranibizumab

SUMMARY:
This is a open label, multicenter, Phase II study to evaluate the usability of the pre-filled syringe (PFS) of SB11 (ranibizumab biosimilar). Healthcare Professionals (HCPs) followed the Instructions for Use (IFU) to prepare and administer SB11 PFS with intravitreal injection to subjects with nAMD or Macular Oedema Secondary to RVO.

DETAILED DESCRIPTION:
This is an open-label, single group, single dose study in subjects with nAMD or Macular Oedema Secondary to RVO.

Screening and Day 1 can be performed on the same day. Subjects will receive ITV injection of SB11 PFS (0.5 mg ranibizumab in 0.05 mL) on Day 1, and follow up visit will be made on Day 1 (+2).

ELIGIBILITY:
Inclusion Criteria:

* Neovascular AMD or macular oedema secondary to RVO in the study eye
* Study eye deemed to be indicated for ranibizumab ITV therapy at the discretion of the ophthalmologist (e.g., retina specialist)
* Aged 18 years and older at the time of signing the informed consent form (ICF)
* Written ICF must be obtained from the subject prior to any study-related procedure (if the subject cannot read ICF, an impartial witness will be present during the entire informed consent discussion)
* Willingness and ability to undertake all scheduled visits and assessments

Exclusion Criteria:

* Best Corrected Visual Acuity (BCVA) of the level of Finger Count or worse [i.e., 0 letter reading using Early Treatment Diabetic Retinopathy Study (ETDRS) chart] in one or both eyes at Screening or at Day 1
* History of and/or current intraocular inflammation (any grading from trace and greater is excluded), including non-infectious uveitis, infectious uveitis, or scleritis, or history of sterile inflammatory reaction after the past ITV injections with any agent in either eye
* Active or suspected infectious disease, or active disorder that preclude safe use of IP at the discretion of the Investigator, in either eye or adnexa of either eye at Screening or at Day 1
* History of excessive bleeding and recurrent haemorrhages, including any prior excessive intraocular bleeding or haemorrhages after ITV injection or intraocular procedures in either eye
* History of massive subconjunctival haemorrhages of concern reported by the subject after an ITV injection in either eye
* Uncontrolled intraocular pressure (IOP) greater than (≥) 25 mmHg in the study eye at Screening or at Day 1
* Treatment with any ITV injection within the 30 days prior to Day 1 in the study eye
* Any invasive ocular surgery including retinal detachment surgery, long-acting ocular therapeutic agent/implant including corticosteroid, or ocular drug release device implant (approved or investigational) in the study eye within 90 days prior to Day 1 or planned intraocular surgery within next 28 days after Day 1
* Ocular laser surgery in study eye at any time within the past 30 days prior to Day 1
* Treatment with any ocular IP in either eye within 90 days prior to Day 1
* Treatment with systemic anti-Vascular Endothelial Growth Factor (anti-VEGF) within 180 days prior to Day 1
* Receipt of any systemic (non-ocular) IP within 180 days prior to Day 1
* Use of therapies that are known to be toxic to ocular tissue within the 180 days prior to Day 1, including, but not limited to, deferoxamine, chloroquine/hydroxychloroquine, tamoxifen, phenothiazines, vigabatrin, or ethambutol
* Known ocular or non-ocular conditions that per the ophthalmologist (e.g., retina specialist) represent a contraindication to ranibizumab use in the patient or may represent an unwarranted patient risk
* Uncontrolled hypertension (defined as systolic blood pressure >160 mmHg and/or diastolic blood pressure >100 mmHg while sitting confirmed after repeated measurement) at Screening or Day 1
* Current systemic infectious disease or therapy for active infectious disease
* Pregnant or lactating women at Screening or at Day 1

Note: Other Protocol Defined Inclusion/Exclusion Criteria Apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-11-21 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Oleksy, M.D., Principal Investigator — Centrum Medyczne Dietla 19 Krakow
Locations (3):
- Poland (3):
  - SB Investigational Site, Katowice
  - SB Investigational Site, Krakow
  - SB Investigational Site, Olsztyn

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee Y, Zalewski D, Oleksy P, Wylegala E, Orski M, Lee J, Kim S. Usability of the SB11 Pre-filled Syringe (PFS) in Patients with Retinal Diseases. Adv Ther. 2024 Aug;41(8):3426-3436. doi: 10.1007/s12325-024-02937-3. Epub 2024 Jul 8. PMID 38976126

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 34 subjects were enrolled for this study and 4 HCPs participated in this study.
Groups:
- SB11 PFS - Subjects: Subjects received a single dose of SB11 PFS containing 0.5 mg ranibizumab in 0.05 mL solution (Day 1).
  4 HCPs participated in this study to administer SB11 PFS to total of 34 subjects.
Period: Overall Study
Arm/Group | SB11 PFS - Subjects
Started | 34
Completed | 34
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 34 subjects were enrolled in the study.
Arm/Group | SB11 PFS
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.1 (7.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 34
  More than one race | 0
  Unknown or Not Reported | 0
Main Indication [Count of Participants; unit: Participants]
  Neovascular AMD | 32
  Macular Oedema Secondary to RVO | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Successful Task Completions
Description: Total of 12 tasks were evaluated, and the percentage of HCP's successful task completions were measured.
  Participating HCPs were allotted sufficient time to review the instructions for use (IFU) before preparing and administering the ITV injection on Day 1. HCP participants did not receive any additional training for the SB11 PFS prior to or during the study.
  "Percentage of successful task completions" was used as the unit of measure, as one SB11 PFS administration procedure is consisted of 12 tasks and the primary endpoint was the percentage of successful tasks completion among total attempts in this study.
Time Frame: Day 1
Population: Overall, 4 participating HCPs performed tasks on 34 enrolled patients (a single PFS ITV injection per patient) leading to a total of "34 attempts" for each tasks in this study.
Measure: Number; unit: Percentage of successful task completion
Units Other Than Participants: attempts
Groups:
- SB11 PFS: HCPs administered a single dose of SB11 PFS containing 0.5 mg ranibizumab in 0.05 mL solution to subjects.
  SB11 PFS: SB11 provided in a pre-filled syringe (PFS) containing 0.5 mg ranibizumab in 0.05 mL for ITV injection
Arm/Group | SB11 PFS
Number analyzed (Participants) | 34
Number analyzed (attempts) | 34
Percentage of successful task completion
  Open the carton | 100
  Remove contents | 100
  Peel the lid off the blister pack | 100
  Carefully remove the PFS from the blister using aseptic technique | 100
  Remove the syringe cap | 100
  Attach a needle | 100
  Remove the needle cap | 100
  Set the dose | 100
  Insert the needle into the injection site | 100
  Press the plunger down to inject the medication | 100
  Remove the needle from the injection site | 100
  Dispose product | 100

2. Secondary Outcome: Percentage of Successful Completion on Critical Tasks
Description: Total of 6 tasks were considered as critical task, and the percentage of HCP's successful completion on critical tasks were evaluated.
  "Percentage of successful task completions" was used as the unit of measure, as one SB11 PFS administration procedure is consisted of 12 tasks and the secondary endpoint was the percentage of successful critical tasks (total of 6) completion among total attempts in this study.
Time Frame: Day 1
Population: as for outcome 1
Measure: Number; unit: Percentage of successful task completion
Units Other Than Participants: attempts
Arm/Group | SB11 PFS
Number analyzed (Participants) | 34
Number analyzed (attempts) | 34
Percentage of successful task completion | 100

3. Secondary Outcome: Percentage of Successful Completion on Essential Tasks
Description: Total of 6 tasks were considered as essential task, and the percentage of HCP's successful completion on essential tasks were evaluated.
  "Percentage of successful task completions" was used as the unit of measure, as one SB11 PFS administration procedure is consisted of 12 tasks and the secondary endpoint was the percentage of successful essential tasks (total of 6) completion among total attempts in this study.
Time Frame: Day 1
Population: as for outcome 1
Measure: Number; unit: Percentage of successful task completion
Units Other Than Participants: attempts
Arm/Group | SB11 PFS
Number analyzed (Participants) | 34
Number analyzed (attempts) | 34
Percentage of successful task completion | 100

ADVERSE EVENTS:
Time Frame: Overall Period (Day 7)
Description: Safety analysis was performed in subjects who received at least one IP during the study period, and all 34 (100.0%) subjects were included.
Arm/Group | SB11 PFS
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 2/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SB11 PFS (N=34)
Ocular discomfort (Eye disorders) | 1 (1)
Ocular hyperaemia (Eye disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-07-05): https://cdn.clinicaltrials.gov/large-docs/63/NCT06176963/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-18): https://cdn.clinicaltrials.gov/large-docs/63/NCT06176963/SAP_001.pdf